CLINICAL TRIAL: NCT06711419
Title: Safety and Efficacy of Caudal Neuroplasty Using Epidural Catheter Combined with (PRF) Versus (PRF) Alone Both Targeting the Dorsal Root Ganglion in Patients with Lumbosacral Radicular Pain
Brief Title: Caudal Neuroplasty Using Epidural Catheter Combined with Pulsed Radiofrequency (versus Pulsed Radiofrequency Alone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Elden Owis Shabaan, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRF vs PRF and neuroplasty
Record Dates: First submitted 2024-11-22; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Disc Herniation
Keywords: Pulsed radio freqency; caudal neuroplasty
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Prolactin-Releasing Hormone; Single Person

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP A (Experimental): Thirty-five patients (to compensate dropouts) will be subjected to Combined caudal neuroplasty using epidural catheter (Perifix® Complete Set 16 G) combined with Pulsed Radiofrequency (PRF) targeting the dorsal root ganglion In patients with lumbosacral radicular pain
  Interventions: Procedure: f caudal neuroplasty using epidural catheter combined with Pulsed Radiofrequency (PRF) versus Pulsed Radiofrequency (PRF) alone
- GROUP B (Experimental): Thirty-five patients (to compensate dropouts) will be subjected to Pulsed Radiofrequency (PRF) alone targeting the dorsal root ganglion In patients with lumbosacral radicular pain
  Interventions: Procedure: f caudal neuroplasty using epidural catheter combined with Pulsed Radiofrequency (PRF) versus Pulsed Radiofrequency (PRF) alone

INTERVENTIONS:
Procedure: f caudal neuroplasty using epidural catheter combined with Pulsed Radiofrequency (PRF) versus Pulsed Radiofrequency (PRF) alone — Fluoroscopic guidance was used in all cases with a C-arm system. The patient was prone with a pillow under the lower abdomen. Anteroposterior (AP) images were taken to identify the target level. The C-arm was angled 15-30° to project the spinous process over the contralateral facet ("scotty dog" view). Skin was infiltrated with lidocaine, and a 22-gauge RF cannula was advanced under fluoroscopy. The tip was positioned in the dorsal-cranial quadrant of the intervertebral foramen on lateral images. PRF was applied with 4 cycles at 42°C for 8 minutes after sensory/motor testing. Injections of lidocaine and triamcinolone followed. In caudal neuroplasty, an epidural catheter was placed using the sacral hiatus as a guide. Fluoroscopy confirmed catheter position. Contrast was injected to confirm spread, and hyaluronidase and lidocaine were administered. Afterward, the catheter was removed.

SUMMARY:
Evaluating the superiority of caudal neuroplasty using epidural catheter (Perifix® Complete Set 16 G) combined with Pulsed Radiofrequency (PRF) versus Pulsed Radiofrequency (PRF) alone targeting the dorsal root ganglion In patients with lumbar radicular pain on pain reduction and quality of life within six months follow up.

DETAILED DESCRIPTION:
Lumbosacral radicular pain (LRP) is a frequently encountered symptom, as the annual prevalence in the general population is reported to be from 9.9% to 25% .Acute lumbosacral radiculopathy is a diffuse disease process that affects more than one underlying nerve root, causing pain, loss of sensation, and motor function depending on the severity of nerve compression. Lumbosacral radiculopathy is very common. Most cases of lumbosacral radiculopathy are self-limited. The most common symptom in radiculopathy is paresthesia.Another common presentation is back pain radiating into the foot, with a positive straight leg raising test. Muscle strength is often preserved in the case of radiculopathy because muscles often receive innervation from multiple roots. Thus, muscle strength is often only affected by severe cases of radiculopathy.[2] The most common causes of lumbar radiculopathy are either a herniated disc with resultant nerve root compression or spondylosis. This process can be acute or can develop chronically over time. Imaging is not always a helpful diagnostic modality as almost 27% of patients without back pain have been found to have disc herniation on magnetic resonance imaging (MRI). Furthermore, this incidental finding does not appear to be predictive of future development of back pain. To diagnose a herniated disc as a source of a patient's pain, it is important to review the complete history and physical and making sure that the symptoms match the imaging results. Patients with lumbar radicular pain often respond to conservative management.

Patients who do not respond to conservative therapies will likely need an MRI for further evaluation and characterization of nerve root involvement, epidural steroid injections and other interventional treatments should be considered [3-5] . When all other treatments have failed, surgery should be considered. Epidural fibrosis may cause chronic radicular lower back pain, negatively affecting patients' quality of life. Adhesions in the epidural space may occur due to surgical or non-surgical causes. Non-surgical causes include annular tear, infection, hematoma, and administration of intrathecal contrast material . Scar tissue may develop in the ventral, dorsal, and lateral regions of the epidural space. Dorsal epidural fibrosis may develop due to surgical hematoma absorption, ventral epidural fibrosis may develop due to disc defects, and lateral epidural fibrosis may develop due to disc defects, facet hypertrophy, and lateral foraminal stenosis . In the neural foramen, epidural veins accompany the nerve roots. Epidural scar tissue causes compression of the veins, which gives rise to edema in the epidural area Stand-alone epidural fibrosis is not a cause of pain. Epidural fibrosis-induced scar tissue fixes the nerve root in one position, causing inflammation of the nerve root. Inflammation causes stretching and compression of the nerve root and increased pain during movement [4](13).

Diagnosis of epidural fibrosis is made by physical examination and radiographic methods, including magnetic resonance imaging (MRI), computed tomography (CT), epidurography, and epidural endoscopy. The gold standard diagnostic method is epidural endoscopy .

Epidural neuroplasty, also known as epidural lysis, can be used to treat epidural fibrosis.

Epidural lysis is commonly performed in patients with radiculopathy and nerve root compression caused by epidural scar tissue. The objective of lysis of adhesion areas in neuroplasty is to deliver the drug to the target areas by opening up the scar tissue in order to suppress inflammation Radiofrequency (RF) procedures have been used to provide long term relief for radicular pain . There are two types of RF procedures: ablative and pulsed. Ablative RF (aRF) requires temperatures of 70-80°C and results in neuronal destruction, Pulsed RF (pRF) is usually deployed at temperatures of 40-45°C, thereby avoiding loss of neuronal function but resulting in presumed neuromodulatory effects that contribute to analgesia, The most commonly used sequence for pRF is a pulse frequency of 2 Hz and a pulse width of 20 milliseconds with the treatment delivered over 2-10 min PRF is believed to have a neuromodulator effect rather than a neurorestorative effect which is particularly advantageous during treatment. PRF is a non-neurolytic lesioning technique for pain palliation, and no proof of neural damage has been reported after PRF administration.

Erdine et al. reported that PRF treatment caused microscopic detriment to the internal ultrastructural components of axons, which leads to the deterioration and disorganization of membrane and mitochondrial morphology and microfilaments and microtubules In this study, a trial seeks to find out the safety efficacy and cost-effectiveness of two different nonoperative approaches in patients with lumbosacral radicular pain short- and long-term outcomes as regards its implications on pain reduction ,analgesic consumption, and the patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 20-80 years old complaining with lumbosacral radicular pain.
* pain intensity ≥4 out of 10 on the numerical rating scale (NRS).
* dominant leg pain with less intense back pain.
* previous failure of conservative management such as physiotherapy, exercise therapy, or analgesic medications.
* Epidural injections administered ≥12 weeks prior to recruitment were permitted because most of the patients visiting our clinic had a history of interlaminar or transforaminal epidural injections.
* Magnetic resonance imaging (MRI) was obtained in all patients and the diagnosis of lumbar disc prolapse was confirmed.

Exclusion Criteria:

* patient refusal to participate in the study,
* age <20 years,
* unbearable pain >9-points on NRS, pain <4-points on NRS.
* signs of progressive motor weakness or neurologic deficits.
* Instability of the spine
* allergies to steroids or contrast dyes.5
* coagulopathy.
* steroid injection within the previous 12 weeks.
* systemic infection, injection site infection.
* malignancy.
* unstable medical or psychiatric condition

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2027-09-10 (Estimated); Study Completion 2028-03-10 (Estimated)

PRIMARY OUTCOMES:
improvement in pain intensity using VAS score | baseline
  The most effective modality in reducing the intensity of pain in patients with lumbar radicular pain

SECONDARY OUTCOMES:
duration of analgesic effect | baseline
  Duration of the analgesic effect following RF procedures

CONTACTS AND LOCATIONS:
Overall Officials: Kilani Ali Abdel-salam, PROF, Study Chair — Assiut University; Saeid Metwally El Sawy, DR, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsao BE, Levin KH, Bodner RA. Comparison of surgical and electrodiagnostic findings in single root lumbosacral radiculopathies. Muscle Nerve. 2003 Jan;27(1):60-4. doi: 10.1002/mus.10291. PMID 12508296
- [Background] Weir BK. Prospective study of 100 lumbosacral discectomies. J Neurosurg. 1979 Mar;50(3):283-9. doi: 10.3171/jns.1979.50.3.0283. PMID 422980
- [Background] van der Windt DA, Simons E, Riphagen II, Ammendolia C, Verhagen AP, Laslett M, Deville W, Deyo RA, Bouter LM, de Vet HC, Aertgeerts B. Physical examination for lumbar radiculopathy due to disc herniation in patients with low-back pain. Cochrane Database Syst Rev. 2010 Feb 17;(2):CD007431. doi: 10.1002/14651858.CD007431.pub2. PMID 20166095
- [Background] Jensen MC, Brant-Zawadzki MN, Obuchowski N, Modic MT, Malkasian D, Ross JS. Magnetic resonance imaging of the lumbar spine in people without back pain. N Engl J Med. 1994 Jul 14;331(2):69-73. doi: 10.1056/NEJM199407143310201. PMID 8208267
- [Background] Boden SD, Davis DO, Dina TS, Patronas NJ, Wiesel SW. Abnormal magnetic-resonance scans of the lumbar spine in asymptomatic subjects. A prospective investigation. J Bone Joint Surg Am. 1990 Mar;72(3):403-8. PMID 2312537
- [Background] Yildirim HU, Akbas M. Percutaneous and Endoscopic Adhesiolysis. Agri. 2021 Jul;33(3):129-141. doi: 10.14744/agri.2020.70037. PMID 34318919
- [Background] Veizi E, Hayek S. Interventional therapies for chronic low back pain. Neuromodulation. 2014 Oct;17 Suppl 2:31-45. doi: 10.1111/ner.12250. PMID 25395115
- [Background] Pushparaj H, Hoydonckx Y, Mittal N, Peng P, Cohen SP, Cao X, Bhatia A. A systematic review and meta-analysis of radiofrequency procedures on innervation to the shoulder joint for relieving chronic pain. Eur J Pain. 2021 May;25(5):986-1011. doi: 10.1002/ejp.1735. Epub 2021 Feb 6. PMID 33471393
- [Background] Van Boxem K, van Bilsen J, de Meij N, Herrler A, Kessels F, Van Zundert J, van Kleef M. Pulsed radiofrequency treatment adjacent to the lumbar dorsal root ganglion for the management of lumbosacral radicular syndrome: a clinical audit. Pain Med. 2011 Sep;12(9):1322-30. doi: 10.1111/j.1526-4637.2011.01202.x. Epub 2011 Aug 3. PMID 21812907